CLINICAL TRIAL: NCT03243474
Title: Non-invasive Monitoring for Early Detection of Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Kardio-Med Silesia (Other)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Principal Investigator, Zbigniew Kalarus, Professor, Kardio-Med Silesia
Other Study IDs: NOMED-AF
Record Dates: First submitted 2017-08-01; First posted 2017-08-09 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 65 - 69 years: The assessment of AF prevalence with use of the monitoring system, blood pressure (BP) measurements and a blood sample collection in patients aged 65 - 69 years.
- 70 - 74 years: The assessment of AF prevalence with use of the monitoring system, blood pressure (BP) measurements and a blood sample collection in patients aged 70 - 74 years
- 75- 79 years: The assessment of AF prevalence with use of the monitoring system, blood pressure (BP) measurements and a blood sample collection in patients aged 75 - 79 years
- 80 - 84 years: The assessment of AF prevalence with use of the monitoring system, blood pressure (BP) measurements and a blood sample collection in patients aged 80 - 84 years
- 85 - 89 years: The assessment of AF prevalence with use of the monitoring system, blood pressure (BP) measurements and a blood sample collection in patients aged 85- 89 years
- ≥90 years: The assessment of AF prevalence with use of the monitoring system, blood pressure (BP) measurements and a blood sample collection in patients aged ≥90 years

SUMMARY:
The aim of this project is to recognize the actual frequency of atrial fibrillation in the Polish population as well as to determine the independent risk factors for the occurrence of its clinically symptomatic and asymptomatic forms

DETAILED DESCRIPTION:
The AF Survey is a cross-sectional observational study aimed to assess the prevalence and control of AF and its correlation with CVD risk factors in Poland, based on a representative sample of adults aged 65+. The main aim of the survey is to assess the prevalence, detectability and control of AF, heart failure, vascular diseases, arterial hypertension, stroke, sedentary lifestyle, smoking, lipid disorders, metabolic syndrome, obesity and diabetes, as well as other factors related to CVD risk such as chronic kidney and liver diseases, sleeping disorders, depression and selected psychosocial factors.

The assessment of AF prevalence with use of the monitoring system developed and validated during the first phase of the project, would be composed of a questionnaire, follow-up data sheet, blood pressure (BP) measurements and a blood sample collection.

The survey consists of three visits to subjects' homes (day: 1; 10+/-4 days and 30+/-4 days) and one phone contact one year after first visit and would be performed by trained nurses. The monitoring system would be installed during the first visit for all patients who sign informed consent form and returned at the third visit one month later. The main questionnaire will be completed during the first visit, which included detailed questions about present health status and history of diseases, hospitalizations, and current medications. The socioeconomic part of the questionnaire included questions concerning the personal and family situation, economic status, household structure, leisure activities, hobbies, and social life. During this visit the Geriatric scale of depression evaluation will be given to the subject to be self-completed, and will be collected at the second visit. BP readings would be taken three times during each visit to the patient's home. Anthropometric measurements are taken twice: at visit one and visit three at the end of the ECG monitoring. Blood samples are taken from subjects at the second visit after 10 to 12-hour fasting. The follow-up data sheet would be completed at the initial visit and at the follow-up visit twelve months after inclusion to the survey. The fieldwork is subcontracted to a company specializing in market research projects for the private and public sectors. The transportation of biological material to the Central Laboratory has been subcontracted to a company with expertise in blood sample transport over long distances. Interviewers will be recruited from among professionally active nurses. Most of them will be social nurses working within local communities. All nurses participating in the survey will complete special training prepared for fieldwork executors of the NOMED-AF project.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 65 years

Exclusion Criteria:

* age < 65 years

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The survey was designed as a country representative study and was carried out on a sample of Polish residents aged ≥65 years, divided into six age groups of equal size and gender proportion (65-69, 70-74, 75-79, 80-84, 85-89 and 90+ years). The planned size of the research sample was 3,000 subjects (250 subjects for each gender and age group). Research participants were randomly recruited in clusters, in a stratified, proportional draw performed in three stages. The reason for overrepresentation of the oldest age groups was to allow separate analysis of data for older people.
Sampling Method: Non-Probability Sample
Enrollment: 3014 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation incidence in general population | 1 year
  the prevalence of atrial fibrillation

SECONDARY OUTCOMES:
Heart failure incidence | 1 year
  the prevalence of heart failure
Stroke incidence | 1 year
  the prevalence of stroke
Atrial hypertension incidence | 1 year
  the prevalence of arterial hypertension
Vascular diseases incidence | 1 year
  the prevalence of vascular diseases

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew Kalarus, Professor, Principal Investigator — KardioMed Silesia
Locations (7):
- Poland (7):
  - Medical University of Gdańsk, Gdansk
  - Jagiellonian University - Medical College, Krakow
  - Pomeranian Medical Uniwersity in Szczecin, Szczecin
  - Comarch Healthcare, Warsaw
  - Medical University of Warsaw, Warsaw
  - Kardio-Med Silesia, Zabrze
  - Institute of Medical Technology and Equipment, Zabrze

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication

REFERENCES:
- [Background] Israel CW, Gronefeld G, Ehrlich JR, Li YG, Hohnloser SH. Long-term risk of recurrent atrial fibrillation as documented by an implantable monitoring device: implications for optimal patient care. J Am Coll Cardiol. 2004 Jan 7;43(1):47-52. doi: 10.1016/j.jacc.2003.08.027. PMID 14715182
- [Background] Lau JK, Lowres N, Neubeck L, Brieger DB, Sy RW, Galloway CD, Albert DE, Freedman SB. iPhone ECG application for community screening to detect silent atrial fibrillation: a novel technology to prevent stroke. Int J Cardiol. 2013 Apr 30;165(1):193-4. doi: 10.1016/j.ijcard.2013.01.220. Epub 2013 Mar 7. No abstract available. PMID 23465249
- [Background] Grond M, Jauss M, Hamann G, Stark E, Veltkamp R, Nabavi D, Horn M, Weimar C, Kohrmann M, Wachter R, Rosin L, Kirchhof P. Improved detection of silent atrial fibrillation using 72-hour Holter ECG in patients with ischemic stroke: a prospective multicenter cohort study. Stroke. 2013 Dec;44(12):3357-64. doi: 10.1161/STROKEAHA.113.001884. Epub 2013 Oct 15. PMID 24130137
- [Background] Glotzer TV, Hellkamp AS, Zimmerman J, Sweeney MO, Yee R, Marinchak R, Cook J, Paraschos A, Love J, Radoslovich G, Lee KL, Lamas GA; MOST Investigators. Atrial high rate episodes detected by pacemaker diagnostics predict death and stroke: report of the Atrial Diagnostics Ancillary Study of the MOde Selection Trial (MOST). Circulation. 2003 Apr 1;107(12):1614-9. doi: 10.1161/01.CIR.0000057981.70380.45. Epub 2003 Mar 24. PMID 12668495
- [Background] Quinn FR, Gladstone D. Screening for undiagnosed atrial fibrillation in the community. Curr Opin Cardiol. 2014 Jan;29(1):28-35. doi: 10.1097/HCO.0000000000000018. PMID 24281348
- [Background] Friberg L, Engdahl J, Frykman V, Svennberg E, Levin LA, Rosenqvist M. Population screening of 75- and 76-year-old men and women for silent atrial fibrillation (STROKESTOP). Europace. 2013 Jan;15(1):135-40. doi: 10.1093/europace/eus217. Epub 2012 Jul 11. PMID 22791299
- [Background] Fernandez V, Bejot Y, Zeller M, Hamblin J, Daubail B, Jacquin A, Maza M, Touzery C, Cottin Y, Giroud M. Silent atrial fibrillation after ischemic stroke or transient ischemic attack: interest of continuous ECG monitoring. Eur Neurol. 2014;71(5-6):313-8. doi: 10.1159/000357561. Epub 2014 Mar 26. PMID 24685765
- [Background] Marfella R, Sasso FC, Siniscalchi M, Cirillo M, Paolisso P, Sardu C, Barbieri M, Rizzo MR, Mauro C, Paolisso G. Brief episodes of silent atrial fibrillation predict clinical vascular brain disease in type 2 diabetic patients. J Am Coll Cardiol. 2013 Aug 6;62(6):525-30. doi: 10.1016/j.jacc.2013.02.091. Epub 2013 May 15. PMID 23684685
- [Background] Cha MJ, Park HE, Lee MH, Cho Y, Choi EK, Oh S. Prevalence of and risk factors for silent ischemic stroke in patients with atrial fibrillation as determined by brain magnetic resonance imaging. Am J Cardiol. 2014 Feb 15;113(4):655-61. doi: 10.1016/j.amjcard.2013.11.011. Epub 2013 Nov 23. PMID 24360776
- [Background] Vermeer SE, Prins ND, den Heijer T, Hofman A, Koudstaal PJ, Breteler MM. Silent brain infarcts and the risk of dementia and cognitive decline. N Engl J Med. 2003 Mar 27;348(13):1215-22. doi: 10.1056/NEJMoa022066. PMID 12660385
- [Background] Camm AJ, Lip GY, De Caterina R, Savelieva I, Atar D, Hohnloser SH, Hindricks G, Kirchhof P; ESC Committee for Practice Guidelines (CPG). 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: an update of the 2010 ESC Guidelines for the management of atrial fibrillation. Developed with the special contribution of the European Heart Rhythm Association. Eur Heart J. 2012 Nov;33(21):2719-47. doi: 10.1093/eurheartj/ehs253. Epub 2012 Aug 24. No abstract available. PMID 22922413
- [Background] Engdahl J, Andersson L, Mirskaya M, Rosenqvist M. Stepwise screening of atrial fibrillation in a 75-year-old population: implications for stroke prevention. Circulation. 2013 Feb 26;127(8):930-7. doi: 10.1161/CIRCULATIONAHA.112.126656. Epub 2013 Jan 23. PMID 23343564
- [Background] Lip GY, Laroche C, Dan GA, Santini M, Kalarus Z, Rasmussen LH, Oliveira MM, Mairesse G, Crijns HJ, Simantirakis E, Atar D, Kirchhof P, Vardas P, Tavazzi L, Maggioni AP. A prospective survey in European Society of Cardiology member countries of atrial fibrillation management: baseline results of EURObservational Research Programme Atrial Fibrillation (EORP-AF) Pilot General Registry. Europace. 2014 Mar;16(3):308-19. doi: 10.1093/europace/eut373. Epub 2013 Dec 17. PMID 24351881
- [Derived] Gumprecht J, Lip GYH, Sokal A, Sredniawa B, Stokwiszewski J, Zdrojewski T, Rutkowski M, Grodzicki T, Kazmierczak J, Opolski G, Kalarus Z. Impact of diabetes mellitus severity, treatment regimen and glycaemic control on atrial fibrillation prevalence in the Polish population aged >/= 65. Sci Rep. 2023 Oct 12;13(1):17252. doi: 10.1038/s41598-023-43939-5. PMID 37828071
- [Derived] Gumprecht J, Lip GYH, Sokal A, Sredniawa B, Mitrega K, Stokwiszewski J, Wierucki L, Rajca A, Rutkowski M, Zdrojewski T, Grodzicki T, Kazmierczak J, Opolski G, Kalarus Z. Relationship between diabetes mellitus and atrial fibrillation prevalence in the Polish population: a report from the Non-invasive Monitoring for Early Detection of Atrial Fibrillation (NOMED-AF) prospective cross-sectional observational study. Cardiovasc Diabetol. 2021 Jun 24;20(1):128. doi: 10.1186/s12933-021-01318-2. PMID 34167520